CLINICAL TRIAL: NCT02414490
Title: Intravenous Immunoglobulin (IVIg) Treatment-Related Fluctuations in Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Patients Using Daily Grip Strength Measurements (GRIPPER)
Brief Title: IVIg Treatment-Related Fluctuations in CIDP Patients Using Daily Grip Strength Measurements
Acronym: GRIPPER
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: BriovaRx Infusion Services (Industry); CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: AHS1-13-001
Record Dates: First submitted 2015-03-13; First posted 2015-04-10 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: CIDP
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood taken for future use will be obtained with each serum IgG sample.

INTERVENTIONS:
Drug: Intravenous Immunoglobulin — The decision to treat with IVIg will be entirely at the discretion of the patient's treating physician.
  Other Names: IVIg

SUMMARY:
This is a prospective observational study of 30 adult CIDP patients who receive home IVIg infusion services from AxelaCare Health Solutions, LLC. The decision to treat with IVIg will be entirely at the discretion of the patient's treating physician.

DETAILED DESCRIPTION:
Subjects will be recruited by individual site investigators. Prior to enrollment each potential subject will have their screening data reviewed by a panel of medical experts for confirmation of inclusion criteria. Each reviewer will be an independent, board-certified, practicing and experienced neurologist with a special interest in CIDP.

Enrolled subjects who have provided informed consent will be instructed to perform and document daily Jamar hand-held Dynamometer grip strength measurements in a paper diary for a 6 month time frame.

Weekly nursing visits will capture disability assessments, physical tests, adverse event and concomitant medications assessment, and other clinical changes that may affect grip strength measurements. Nurses will review each subjects captured grip data from paper diary on an iPad during weekly home assessments. Nurses will also administer the HRQOL Short-Form (SF) 36 questionnaire at the baseline, week 12 and week 24 study visits.

Serum immunoglobulin G (IgG) levels will be captured by the home study nurse at three time points surrounding IVIg infusions and will be classified as either trough, peak, or mid. Each subject will have serum Ig collected by blood draw for the first 4 IVIg treatment cycles, for a total of 12 blood draws per subject.

The "trough" serum IgG level will be collected immediately prior to Ig infusion. The "peak" serum IgG level will be collected 5 minutes post-Ig infusion. The "mid" serum IgG level will be collected two weeks post-Ig infusion.

There are currently no known biomarkers that can assist with CIDP diagnosis, prognosis, or treatment optimization. As part of this study, subjects will be required to have additional blood taken and stored for future use. Future use may include the possible discovery of specific biomarkers predicting the response to IVIg or other therapies, optimization of IVIg dosage based on pharmacodynamics, pathogenesis of CIDP, and more effective CIDP diagnostic markers. Blood taken for future use will be obtained with each serum IgG sample. No additional blood draws will be required.

Should IVIg therapy be discontinued during the study, daily grip strength measurements will continue to be performed and recorded in the subject diary for up to 30 days or to the end of the study, whichever comes first. Weekly nurse visits with collection of the disability assessments and serum IgG blood draws will continue for up to 4 home nurse visits or until the end of the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Definite or probable CIDP according to the European Federation of Neurological Studies (ENFS)/Peripheral Nerve Society (PNS) criteria 2010
2. Inflammatory Neuropathy Cause and Treatment Group (INCAT) upper limb disability score of 2 or greater at any time during disease
3. CIDP Disease Activity Status (CDAS) classification of Stable Active Disease or Improvement at time of screening
4. Men or women age 18-85 years
5. Receiving physician prescribed intravenous immunoglobulin (IVIg) therapy with a treatment interval between a minimum of 21 days and a maximum of 42 days
6. Be on a stable dose of IVIg for at least 3 months prior to study participation
7. With proper training from a healthcare professional, demonstrate proficiency in the ability to perform daily Jamar Dynamometer grip strength measurements
8. Ability to have an adult present (e.g., spouse, adult child) to assist with daily Dynamometer grip strength measurement, if needed
9. Eligible for infusion services by AxelaCare Health Solutions, LLC, in collaboration with the subject's prescribing physician and insurance provider
10. Ability to read and write English
11. Ability and willingness to provide informed consent and comply with study requirements and procedures
12. Confirmation of diagnosis of CIDP by outside expert panel

Exclusion Criteria:

1. Any polyneuropathy of other causes, including multifocal motor neuropathy, hereditary demyelinating neuropathy, POEMS syndrome, polyneuropathy associated with diabetes mellitus, polyneuropathy associated with systemic lupus erythematosus
2. Subjects who, by majority vote of the outside expert panel do not meet diagnostic criteria for CIDP or probably CIDP
3. CDAS classification of Cure, Remission, or Unstable Active Disease
4. The presence of any type of recent arm and/or hand bone fracture
5. The presence of any medical condition that the investigator and/or prescribing physician deems incompatible with participation in this trial
6. Receiving subcutaneous immunoglobulin (SCIg) therapy during study participation
7. Receiving pulse dose corticosteroids during study participation (daily corticosteroids are allowed provided dose equal or less than prednisone 20 mg daily and no anticipated dose changes during the study)
8. Prisoners
9. Ward of the state

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include men and women between 18-85 years of age currently being treated with IVIg. Up to 30 subjects with a definite or probable diagnosis of CIDP as defined by the EFNS/PNS criteria and confirmed by outside review will be enrolled.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Daily grip strength (GS) measurements | 6 months
  Extent of treatment related fluctuations to intravenous immunoglobulin (IVIg) in patients with Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) using a Jamar Dynamometer to capture daily grip strength (GS) measurements

SECONDARY OUTCOMES:
Percentage of IVIg treatment cycles in which the maximum and minimum grip strength (GS) measurements differ by more than 10% of the maximum | 6 months
  Determine the percentage of IVIg treatment cycles in which the maximum and minimum grip strength (GS) measurements differ by more than 10% of the maximum and determine the percentage of subjects who have fluctuations of that magnitude.
Rasch-built Overall Disability Scale | 6 months
  Changes in Rasch-built Overall Disability Scale in the event a treating physician decides to modify IVIg therapy during study participation.
Timed Up and Go test | 6 months
  Changes in Timed up and Go test in the event a treating physician decides to modify IVIg therapy during study participation.
Overall Neuropathy Limitations Scale | 6 months
  Changes in Overall Neuropathy Limitations Scale in the event a treating physician decides to modify IVIg therapy during study participation.
Health-Related Quality of Life (HRQOL) | 6 months
  Changes in Health-Related Quality of Life (HRQOL) at three time points during the study (baseline, Week 12 and Week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Allen, MD, Principal Investigator — University of Minnesota
Locations (7):
- United States (7):
  - Neurology at John's Creek, Johns Creek, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center/Dartmouth Geisel School of Medicine, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Allen JA, Pasnoor M, Dimachkie MM, Ajroud-Driss S, Brannagan TH, Cook AA, Walton T, Fiecas MB, Kissel JT, Merkies I, Gorson KC, Lewis RA. Quantifying Treatment-Related Fluctuations in CIDP: Results of the GRIPPER Study. Neurology. 2021 Apr 6;96(14):e1876-e1886. doi: 10.1212/WNL.0000000000011703. Epub 2021 Feb 16. PMID 33593867